CLINICAL TRIAL: NCT03213444
Title: Impact of Adjuvant Chemotherapy in Cardiovascular Autonomic Regulation in Patients With Colon Cancer
Brief Title: Impact of Adjuvant Chemotherapy in Patients With Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant Chemotherapy
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2016-07

CONDITIONS: Colon Cancer; Adjuvant Chemotherapy
Keywords: Colon cancer; adjuvant chemotherapy; sympathetic nerve activity; peripheral vascular function
MeSH Terms: conditions — Colonic Neoplasms | interventions — Chemotherapy, Adjuvant; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Patients with stage II disease undergoing adjuvant 5-FU treatment will be allocat in chemotherapy-1 group, while stage III patients undergoing combined adjuvant chemotherapy (5FU + Oxaliplatin) will be allocat to the Chemotherapy group -2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quimioterapy 1 (Active Comparator): adjuvant chemotherapy with 5-FU isolated
  Interventions: Drug: adjuvant chemotherapy with 5-FU isolated
- Quimioterapy 2 (Active Comparator): adjuvant chemotherapy with 5-FU associated with oxaliplatin
  Interventions: Drug: adjuvant chemotherapy with 5-FU associated with oxaliplatin

INTERVENTIONS:
Drug: adjuvant chemotherapy with 5-FU isolated — Patients submitted to adjuvant chemotherapy with 5-FU isolated
  Arms: Quimioterapy 1
Drug: adjuvant chemotherapy with 5-FU associated with oxaliplatin — Patients submitted to adjuvant chemotherapy with 5-FU associated with oxaliplatin
  Arms: Quimioterapy 2

SUMMARY:
The present study aims to investigate the impact of adjuvant chemotherapy with 5-FU isolated and associated with oxaliplatin in cardiac autonomic control and endothelium-dependent vascular function in patients undergoing colectomy for stages II and III colon cancer. Will be performed evaluation of cardiac and vascular function, autonomic control, functional capacity and blood evaluations.

DETAILED DESCRIPTION:
Cancer is a major public health problem. Colorectal cancer is the third most common cancer in men and women around the world. Despite advances in surgical and pharmacological treatment, this type of cancer remains a leading cause of cancer death in Western countries. The adjuvant chemotherapy treatment based on the use of fluoropyrimidine, especially 5-fluorouracil (5-FU) is the mainstay of the pharmacological treatment of colorectal cancer. This treatment showed benefit in overall survival and progression-free survival in the adjuvant treatment of patients with stage II and III disease. In the last decade, the combination treatment with oxaliplatin has shown benefit in patients with either metastatic disease as with locoregional disease who underwent surgical treatment. However, the increased use of 5-FU and oxaliplatin, and increased patient survival have caused increased incidence of adverse events. 5-FU has cardiotoxic effects that may range from 1.2 to 18% depending upon the drug administration. Another adverse event of chemotherapy for colon cancer is neurotoxicity. Peripheral neuropathy is one of the toxicities associated with treatment with Oxaliplatin and its characteristics to be dose-dependent and cumulative. Thus, the adjuvant chemotherapy with 5-FU and oxaliplatin may cause cardiotoxicity, changes in vascular function and increased oxidative stress. What is not known are the effects of treatment of 5-FU and oxaliplatin in cardiac autonomic modulation and peripheral vascular function. Therefore, the present study aims to investigate the impact of adjuvant chemotherapy with 5-FU isolated and associated with oxaliplatin in cardiac autonomic control and endothelium-dependent vascular function in patients undergoing colectomy for stages II and III colon cancer. Will be performed evaluation of cardiac and vascular function, autonomic control, functional capacity and blood evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Scale of Performance Status 0 - 1
* Patients submitted to colectomy for adenocarcinoma of colon stages II and III.

Exclusion Criteria:

* Severe pulmonary disease
* Decompensated cardiovascular disease
* Neurological disease
* Insulin-dependent diabetes mellitus
* Dialysis renal insufficiency

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
cardiac function evaluation | Change from Baseline cardiac function at 6 months
  Cardiac function will be assessed by two-dimensional (B-mode) echocardiography, pulsed Doppler

SECONDARY OUTCOMES:
vascular function evaluation | Change from Baseline vascular function at 6 months
  Vascular function will be assessed by high resolution Doppler ultrasound
autonomic control evaluation | Change from autonomic control at 6 months
  autonomic control will be assessed by microneurography and heart rate variability
functional capacity evaluation | Change from Baseline functional capacity at 6 months
  functional capacity will be assessed by cardiopulmonary exercise test
Proinflammatory cytokines | Change from Baseline Proinflammatory cytokines at 6 months
  Proinflammatory cytokines will be assessed by blood evaluations

CONTACTS AND LOCATIONS:
Locations (1):
- Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No